CLINICAL TRIAL: NCT04681820
Title: Evaluating Efficacy and Safety of Flumatinib for Chronic Phase Chronic Myeloid Leukemia(CML-CP) Without Optimal Response (Warning or Failure) to Imatinib or Dasatinib: A Prospective, Multicenter, Pragmatic Clinical Trial
Brief Title: Evaluating Efficacy and Safety of Flumatinib for Chronic Phase Chronic Myeloid Leukemia(CML-CP) Without Optimal Response (Warning,Failure) to Imatinib or Dasatinib
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Weiming Li, chief physician, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: HS-2020-07WH
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: CML-CP; Mutation;Suboptimal Response or Failure in TKI
MeSH Terms: interventions — flumatinib; nilotinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- flumatinib: flumatinib 600mg QD, fasting administration
  Interventions: Drug: Flumatinib; Drug: Nilotinib
- nilotinib: nilotinib 400mg BID, fasting administration
  Interventions: Drug: Flumatinib; Drug: Nilotinib

INTERVENTIONS:
Drug: Flumatinib — Flumatinib mesylate tablets 600mg qd for 24 months
Drug: Nilotinib — Nilotinib Capsules 400mg bid for 24 months

SUMMARY:
Imatinib has revolutionized the treatment of chronic myeloid leukemia (CML) and is the current standard of care in the treatment of patients with newly diagnosed CML. However, about 30% of patients still show drug resistance or disease progression. Currently, the most widely studied mechanism of TKI resistance in CML patients is mutations in the ABL kinase region. So far, more than 100 kinase domain mutations have been found in disease progression and imatinib resistance. It is estimated that more than 25% of CML patients will change TKI at least once in their lifetime due to drug resistance or intolerance. The 2020 edition of the "Guidelines for the Diagnosis and Treatment of Chronic Myelogenous Leukemia in China" proposes that patients with F317L/V/I/C, V299L and T315A mutations are more likely to obtain clinical efficacy by switching to the second-generation TKI nilotinib; patients with Y253H, E255K/V and F359C/V/I mutations are more likely to obtain clinical efficacy by switching to the second-generation TKI dasatinib; patients with T315I mutations are resistant to both nilotinib and dasatinib. Flumatinib has been shown to be a more potent inhibitor of BCR-ABL1 tyrosine kinase than imatinib. In vitro studies, it has shown that flumatinib inhibits wild-type and common BCR-ABL mutations(Q252H, V299L, F317L/I, M351T, H396P, etc.) more potently, and the anti-mutation spectrum of flumatinib is similar to nilotinib. Therefore, this study is designed to provide clearer guidance for patients with suboptimal response or failure in the treatment of TKI as well as those who have specific ABL kinase domain mutations during CML treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥18 years of age;
2. CML-CP patients when enrolled

   Definition of diagnosis:

   Bone marrow cytogenetic confirmation of Philadelphia chromosome of t (9;22) translocations and/or the presence of P210 BCR-ABL1 transcripts via molecular assessment;

   Documented chronic phase CML will meet all the criteria defined as:

   < 15% blasts in peripheral blood and bone marrow < 30% blasts plus promyelocytes in peripheral blood and bone marrow < 20% basophils in the peripheral blood

   ≥ 100 x 109/L (≥ 100,000/mm3) platelets No evidence of extramedullary leukemic involvement, with the exception of hepatosplenomegaly
3. CML-CP patients without optimal response(warning or failure) when treated with imatinib or dasatinib.
4. Female patients of childbearing potential must have a negative serum pregnancy test;
5. Ability to provide written informed consent prior to any study related screening procedures being performed.

Exclusion Criteria:

1. Treatment with other tyrosine kinase inhibitor(s) except imatinib and dasatinib prior to study entry;
2. With any mutations as follows :T315I、Y253F/H、E255K/V、F359C/V/I (if there are any other mutations,at physicians' discretion );
3. Entry into another therapeutic clinical trial;
4. Concomitant diseases that, according to the investigator's judgment, pose a serious risk to the patient's safety or completion of the study;
5. History of neurological or psychiatric disorders, including epilepsy or dementia;
6. Major surgery within 4 weeks prior to Day 1 of study;
7. Patients with another primary malignancy,unless the other primary malignancy is currently stable or does not need active intervention;
8. Women of reproductive age or men who are unable to use adequate methods of contraception, including women who are pregnant or breastfeeding;
9. ECOG≥3;
10. Patients who are unable to compliance with study or follow-up procedures;
11. Allergic to any of the components in this trial;
12. Not appropriate to attend this trial judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CML-CP patients without optimal response(warning or failure) treated with imatinib or dasatinib
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Major molecular response rate at 12 months | 12 months
  Major molecular response is defined as ≤ 0.1% BCR-ABL/ABL% by international scale

CONTACTS AND LOCATIONS:
Locations (1):
- Weiming Li, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No